CLINICAL TRIAL: NCT06065059
Title: Phase 1/2, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of TNG348 Single Agent and in Combination With a PARP Inhibitor in Patients With BRCA 1/2 Mutant or Other HRD+ Solid Tumors
Brief Title: Study to Evaluate TNG348 Alone and With a PARP Inhibitor in Patients With BRCA 1/2 Mutant or HRD+ Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to safety
Sponsor: Tango Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG348-C101
Record Dates: First submitted 2023-09-15; First posted 2023-10-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Ovarian Cancer; Pancreas Cancer; Prostate Cancer; BRCA1 Mutation; BRCA-Mutated Ovarian Carcinoma; BRCA-Associated Breast Carcinoma; HRD Positive Advanced Ovarian Cancer
Keywords: BRCA mutant; HRD positive; solid tumors; USP1; TNG348
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: Phase 1 Dose Escalation and Phase 2 Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Single Agent Dose Escalation (Experimental): Participants with BRCA 1/2 mutant or HRD+ solid tumors will receive escalating doses of TNG348 to estimate the MTD
  Interventions: Drug: TNG348
- Combination Dose Escalation (Experimental): Participants with BRCA 1/2 mutant or HRD+ solid tumors will receive escalating doses of TNG348 in combination with olaparib to estimate the MTD
  Interventions: Drug: TNG348; Drug: Olaparib
- Single agent dose expansion in breast cancer (Experimental): Participants with BRCA 1/2 mutant breast cancer will receive TNG348 at the identified RP2D
  Interventions: Drug: TNG348
- Single agent dose expansion in ovarian cancer (Experimental): Participants with BRCA 1/2 mutant ovarian cancer will receive TNG348 at the identified RP2D
  Interventions: Drug: TNG348
- Combination therapy dose expansion in breast cancer (Experimental): Participants with BRCA 1/2 mutant breast cancer will receive TNG348 in combination with olaparib at the identified RP2D
  Interventions: Drug: TNG348; Drug: Olaparib
- Combination therapy dose expansion in ovarian cancer (Experimental): Participants with BRCA 1/2 mutant ovarian cancer will receive TNG348 in combination with olaparib at the identified RP2D
  Interventions: Drug: TNG348; Drug: Olaparib
- Combination therapy dose expansion in pancreatic or prostate cancer (Experimental): Participants with BRCA 1/2 mutant pancreatic or prostate cancer will receive TNG348 in combination with olaparib at the identified RP2D
  Interventions: Drug: TNG348; Drug: Olaparib
- Combination therapy dose expansion in HRD+ advanced or metastatic solid tumors (Experimental): Participants with HRD+ advanced or metastatic solid tumors will receive TNG348 in combination with olaparib at the identified RP2D
  Interventions: Drug: TNG348; Drug: Olaparib

INTERVENTIONS:
Drug: TNG348 — Ubiquitin Specific Peptidase 1 (USP1) inhibitor
Drug: Olaparib — PARP inhibitor
  Other Names: Lynparza
  Arms: Combination Dose Escalation; Combination therapy dose expansion in HRD+ advanced or metastatic solid tumors; Combination therapy dose expansion in breast cancer; Combination therapy dose expansion in ovarian cancer; Combination therapy dose expansion in pancreatic or prostate cancer

SUMMARY:
The goal of this interventional clinical trial is to learn about TNG348, a ubiquitin specific peptidase 1 (USP1) inhibitor, alone and in combination with olaparib in patients with BRCA 1/2 mutant or HRD+ solid tumors.

The main question[s] it aims to answer are:

* to evaluate the safety and tolerability of single agent and combination therapy
* to determine the recommended dose for Phase 2 of single agent and combination therapy
* to determine the pharmacokinetics of TNG348 as a single agent and in combination therapy
* to evaluate the initial antineoplastic activity as a single agent and in combination therapy

Participants will receive study treatment until they experience an undesirable side effect, their disease progresses or until they withdraw consent.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1/2, open-label, multi-center, dose-escalation and expansion study designed to determine the maximum-tolerated dose (MTD) and recommended Phase 2 dose(s) (RP2D) and evaluate the safety, tolerability, and preliminary antitumor activity of TNG348 single agent and in combination with olaparib in participants with BRCA1/2 mutant or other HRD+ advanced or metastatic solid tumors.

In Phase 1 (dose escalation), the single agent component will explore escalating oral doses of TNG348 administered alone and in combination with olaparib.

Participants in Phase 2 (dose expansion) will be dosed at the RP2D(s) determined from Phase 1 based on safety and tolerability demonstrated, along with the available PK data and studied during Phase 1, as applicable.

In the Phase 2 portion of the study, both single agent and combination therapy may be evaluated to assess an early signal of clinical benefit, as well as for confirmation of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years of age at the time of signature of the main study ICF.
* Has ECOG performance status of 0 or 1.
* Has advanced or metastatic solid tumor with measurable disease based on RECIST v1.1.
* All participants must have documented BRCA 1/2 mutant or other HRD+ in solid tumor, which is identified through a validated sequencing test
* Adequate organ and bone marrow function per local labs
* Negative serum pregnancy test result at screening
* Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to TNG348, olaparib or its excipients
* Uncontrolled intercurrent illness that will limit compliance with the study requirements
* Currently participating in or has planned participation in a study of another investigational agent or device
* Impairment of GI function or disease that may significantly alter the absorption of study drug
* Active prior or concurrent malignancy.
* Central nervous system metastases associated with progressive neurological symptoms
* Participant with MDS
* Clinically relevant cardiovascular disease
* Participant with known active or chronic infection
* A female patient who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
To determine dosing for TNG348 alone and in combination (Phase 1 only) | 21 days
  • To determine the MTD, RP2D(s), and dosing schedule of TNG348 single agent and in combination with olaparib
Measure anti-tumor activity using RECIST 1.1 (Phase 2 only) | 56 days
  To assess the antitumor activity of TNG348 single agent and in combination using RECIST 1.1 per investigator assessment

SECONDARY OUTCOMES:
Measure anti-tumor activity using RECIST 1.1 (Phase 1 only) | 56 days
  To assess the antitumor activity of TNG348 single agent and in combination using RECIST 1.1 per investigator assessment
Characterize the safety and tolerability profile | 21 days
  Measure frequency, severity, timing, and relationship to study treatment of any AEs, SAEs, and changes in safety laboratory tests
Characterize the plasma PK profile | 16 days
  To determine the Cmax of TNG348
Characterize the plasma PK profile | 16 days
  To determine the Tmax
Characterize the plasma PK profile | 16 days
  To determine the AUC0-t and AUC0-∞ of TNG348
Characterize the plasma PK profile | 16 days
  To determine the half-life of TNG348
Characterize olaparib concentrations when administered with TNG348 | 16 days
  To characterize the pre treatment and trough concentration levels of olaparib when administered in combination with TNG348
Assess changes in levels of ubPCNA in response to TNG348 as single agent or in combination | 22 days
  Measure ubPCNA in tumor tissue and blood, on study treatment relative to pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Crystal, MD, PhD, Study Director — Tango Therapeutics, Inc.
Locations (7):
- United States (7):
  - HealthONE, Denver, Colorado
  - Mid Florida Cancer Centers, Orange City, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - New York University Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No